CLINICAL TRIAL: NCT00549367
Title: The Role of Diet Education and Nutritional Counselling in the Ongoing Care of People Living With HIV in Thailand (TACH001)
Brief Title: The Role of Diet Education and Nutritional Counselling in the Ongoing Care of People Living With HIV in Thailand
Acronym: TACH001
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thai Red Cross AIDS Research Centre (Other)
Collaborators: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: TACHIN001
Record Dates: First submitted 2007-10-23; First posted 2007-10-25 (Estimated); Last update posted 2023-02-17 (Actual); Status verified 2021-07

CONDITIONS: HIV Infections
Keywords: Nutritional status; Nutrition counselling; Nutrition assessment; HIV; Alternative Medicine; Complementary Medicine
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other): Clients in the control arm of the study will receive nutrition assessment only for the first 24 weeks and the be transferred to nutrition counselling group
  Interventions: Behavioral: Nutrition Counselling

INTERVENTIONS:
Behavioral: Nutrition Counselling — Clients will receive ongoing nutrition assessment and dietary counselling. The intervention arm will receive all baseline assessments and individual nutritional assessment, counselling and nutrition management plans using standards of practice

SUMMARY:
To evaluate the effectiveness of nutrition education and dietary counselling to improve the nutritional status, well-being and quality of life of people living with HIV/AIDS (PLWHA) attending an HIV treatment facility in Bangkok Thailand.

DETAILED DESCRIPTION:
To evaluate the effectiveness of nutrition education and dietary counselling to improve the nutritional status, well-being and quality of life of people living with HIV/AIDS (PLWHA) attending an HIV treatment facility in Bangkok Thailand. This will be achieved by determining if dietary counselling and nutrition education has an effect on nutritional status (weight, lean body mass and fat mass), dietary intake, food security, quality of life, biochemical parameters (including total cholesterol, LDL/ HDL cholesterol and Triglyceride), experience of symptoms and patient satisfaction

ELIGIBILITY:
Inclusion Criteria:

* HIV positive
* 18 years of age or older
* Receiving ongoing care as part of the TRCARC Family Clinic (TRCARC Wellness Plus clinic)
* Either ART naive or have been on stable ART for more than 6 months

Exclusion Criteria:

* HIV negative
* Unintentional weight loss of more than 10% usual body weight, or BMI<17
* BMI>30
* Suspected or documented HIV related opportunistic infection
* Pregnant women
* Women less than 3 months post-partum

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2007-11 (Actual); Primary Completion 2022-12 (Actual); Study Completion 2023-02 (Actual)

PRIMARY OUTCOMES:
body composition measured by BIA and anthropometry | 48 weeks

SECONDARY OUTCOMES:
Change in dietary intake, food security, quality of life, biochemical parameters (including total cholesterol, LDL/ HDL cholesterol and Triglyceride), experience of symptoms and patient satisfaction | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Simon J Sadler, Principal Investigator — Albion Street Centre
Locations (1):
- Thai Red Cross AIDS Research Centre, Bangkok, Pathumwan, Thailand